CLINICAL TRIAL: NCT06270329
Title: Comparison of the Effectiveness of Neuromuscular Training Program and Conventional Physical Therapy Program in Patients With Knee Osteoarthritis.
Brief Title: Neuromuscular Training Program in Patients With Knee OA (Osteoarthritis)
Acronym: OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Eda Ozge OKUR, Asst. Prof., Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMTwithKOA
Record Dates: First submitted 2024-02-10; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
Keywords: Neuromuscular training; Knee osteoarthritis; Physical therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neuromuscular training program (Experimental): Participants were administered the neuromuscular training program 60 min a day, 2 days a week for 8 weeks.
  Interventions: Other: Neuromuscular training program
- conventional physical therapy program (Active Comparator): Participants were administered the conventional physiotherapy program 60 min a day, 2 days a week for 8 weeks.
  Interventions: Other: conventional physical therapy program

INTERVENTIONS:
Other: Neuromuscular training program — Hotpack application TENS (transcutaneous electrical stimulation) Warm-up phase: bicycle ergometer (ten minutes)
  Exercise phase:
  core stabilization and postural control exercises postural orientation exercises lower extremity strengthening exercises functional exercises (balance and proprioception exercises using a balance board) Cool-down Phase
  Arms: neuromuscular training program
Other: conventional physical therapy program — Hotpack application TENS (transcutaneous electrical stimulation) Conventional physical therapy exercises (straight leg raises, knee flexor and extensor strengthening, hip muscle strengthening)
  Arms: conventional physical therapy program

SUMMARY:
The aim of this study was to compare the effects of neuromuscular training program and conventional physical therapy program on pain, functional status, physical performance, balance, muscle strength and quality of life in patients with knee osteoarthritis (KOA).

DETAILED DESCRIPTION:
The study was carried out in Afyonkarahisar Health Sciences University Health Application Research Center in individuals with 2nd or 3rd degree KOA according to Kellgren and Lawrence Classification. The study was planned as a randomized controlled clinical trial design. The study group were recruited to the neuromuscular training program and the control group were recruited to the conventional physical therapy program 5 days a week for 3 weeks. Individuals were evaluated at the baseline and after training programs. Demographic and clinical data were first recorded in the evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Having grade 2 or 3 osteoarthritis according to the Kellgren and Lawrence Classification
* Having pain score of 2 or above on VAS
* Not having received physical therapy in the last 3 months
* Not having received an intra-articular corticosteroid injection in the last 6 months
* Not having used oral corticosteroids in the last month
* Being between the ages of 40-80
* Body mass index being between 19-40 kg/cm2

Exclusion Criteria:

* Systemic arthritis
* Hypertensive condition that prevents exercise
* Pregnancy, cognitive impairment, parkinson-like neurological disorders
* Having had a knee or hip joint replacement

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | At first and third week
  Pain evaluation. The participant is asked to give a score between 1 and 10 for her pain.
Western Ontario and McMasterUniversities Osteoarhritis Index | At first and third week
  Functional status evaluation. The scale consists of 3 subheadings that evaluate pain, stiffness and physical function.
  High Western Ontario and McMasterUniversities Osteoarhritis Index score indicates increased pain and stiffness and deterioration in physical function.
Time on One Leg Standing | At first and third week
  Balance evaluation. Participants were asked to stand on one leg with their eyes open for as long as possible, and the time was measured with a stopwatch and recorded in seconds.
Five Times Sit to Stand Test | At first and third week
  Physical performance evaluation. The time it takes for the patient to sit and stand up from a chair five times is recorded. As time decreases, it indicates better performance.
Manual Muscle Test | At first and third week
  Muscle strength evaluation. A score between 0 and 5 is given depending on muscle strength.
Short Form | At first and third week
  Quality of life evaluation. It consists of 8 subheadings: physical function, problems caused by physical problems, emotional well-being, problems caused by emotional problems, general health, social function, pain, energy/fatigue.
  High scores indicate good health, low scores indicate poor health.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.